CLINICAL TRIAL: NCT01391247
Title: Validation of Retinal Oximetry in Glaucoma Patients: a Structural and Functional Correlation
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S52610
Record Dates: First submitted 2011-06-28; First posted 2011-07-11 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2010-12

CONDITIONS: Open Angle Glaucoma; Low Tension Glaucoma
Keywords: open angle glaucoma; low tension glaucoma; oximetry
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- healthy age machted controls
- normal tension glaucoma patients
- primary open angle glaucoma patients

SUMMARY:
Retinal ischemia is thought to play an important role in the pathogenesis of glaucoma. Up until today, very little is known about the metabolic alterations in the retina of glaucoma patients, since only techniques for surrogate measurements of metabolism (like blood flow velocities and vessel diameter) were available. Oximetry has provided us with an important tool to study metabolism in glaucoma, and to correlate these findings with the available blood flow evaluation techniques. Preliminary results by the group of Prof Stefánsson (2011) with the dual wavelength oximeter pointed out that deeper glaucomatous visual field defects are associated with decreased arteriovenous differences in retinal oxygen saturation. These data suggest that a change in oxygen metabolism occurs in glaucomatous retina. This reduced oxygen metabolism may be related to tissue atrophy. However, this explanation is still hypothetical, since the relation between these oximetry results and structural changes in the optic nerve have not been studied yet.

1. What are the oximetry values in a normal population of within the same age group as the glaucoma population? To answer this question, a normative database of the investigators retinal oximetry device needs to be constructed for healthy controls.
2. Do glaucoma patients have different retinal oximetry values than these normal patients? Are there any differences in retinal oxygenation between these glaucoma groups? To answer these questions, oximetry measurements will be performed in patients with normal tension glaucoma (NTG) and primary open angle glaucoma (POAG).
3. Is there an association between structural optic disc and retinal nerve fibre layer changes, using Heidelberg Retinal Tomography (HRT), with alterations in retinal vascular oxygen saturation in NTG and POAG patients?
4. Are blood flow measurements, using colour Doppler imaging (CDI), correlated with alteration in retinal vascular oxygen in NTG and POAG patients?

DETAILED DESCRIPTION:
1. Oximetry pictures will be taken and analysed.
2. CDI exam will be performed.
3. Visual field examen will be performed.
4. HRT will be performed.

ELIGIBILITY:
Inclusion Criteria:

* individuals over 18 years old
* willing to sign an informed consent and able to comply with the requirements of the study
* having no other ocular diseases besides glaucoma

Exclusion Criteria:

* history of ocular trauma
* intraocular surgery (except for cataract surgery)
* eye disease (except glaucoma)
* systemic diseases with ocular involvement like diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Comparison of oxygen saturation between glaucoma patients and healthy controls. | patients will be followed during their hospital stay, an average. of 3 hours
  Retinal oximetry gives us oxygen saturation values who will be compared between glaucoma patients and healthy controls and will be correlated to visual field mean defect, structure parameters from the HRT and velocity measurements with the CDI.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, Phd, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Department of Ophthalmology, UZLeuven, Leuven, Belgium